CLINICAL TRIAL: NCT06227000
Title: Living Longer and Stronger With Spinal Cord Injury: An Online Program for Promoting Healthy Aging
Brief Title: Living Longer and Stronger With Spinal Cord Injury (SCI)
Acronym: LLS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susan Robinson-Whelen, Adjunct Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MH-23-0383; 90SIMS0019-01-00 (Other Grant/Funding Number: Administration for Community Living)
Record Dates: First submitted 2024-01-16; First posted 2024-01-26 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; aging; health promotion; intervention; randomized controlled trial
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Living Longer and Stronger (LLS) intervention (Experimental)
  Interventions: Behavioral: Living Longer and Stronger with SCI
- Control Group (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Living Longer and Stronger with SCI — Study staff will schedule a brief zoom training session with each person assigned to the intervention to ensure that they are able to download and use the Zoom platform. Once a weekly session day and time has been determined the 8-week LLS intervention program will begin. LLS group participants will participate in 2-hour weekly sessions co-facilitated by a study investigator and one of the study's senior advisors. Participants will be encouraged to set a health-oriented goal and complete weekly action plans. They will be provided with materials each week with health-related information and resources. Participants will also be asked to complete a short survey each week to rate the session. After completing the 8 sessions, a link to the post-test survey and some questions to evaluate the LLS program will be sent to the participants. Finally there will be follow up survey to be completed at 4 months post intervention.
  Arms: Living Longer and Stronger (LLS) intervention
Behavioral: Control — Participants will be sent links to the three surveys at the same time as those assigned to the LLS group but they will not attend any of the zoom calls. They will be offered all study materials at the end of the study.
  Arms: Control Group

SUMMARY:
The purpose of this study is to develop a health promotion group intervention to meet the unique health promotion needs of people aging with SCI, to test the efficacy of the adapted intervention program, Living Longer and Stronger with SCI, in a randomized controlled trial and to assess the mechanisms through which the intervention may enhance physical, psychological, and social health.

ELIGIBILITY:
Inclusion Criteria:

* traumatic spinal cord injury (SCI)
* have traumatic SCI for at least 15 years OR be over the age of 45
* use a manual or power wheelchair for mobility at least some of the time
* reside in the U.S.
* speak and read English
* access to a smart phone, tablet, or a computer with Internet access
* have or be willing to obtain email for study correspondence

Exclusion Criteria:

* cognitive impairment that significantly limits their ability to give informed consent, participate in the intervention, or complete study assessments as determined by an inability to correctly answer questions demonstrating study comprehension
* have a significant visual or hearing impairment that would prohibit their ability to participate in the interactive online intervention with accommodations
* report active suicidality or significant problems with alcohol or other drug use
* live in an institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in physical health as assessed by the SF-36 General Health Subscale | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  a 5-item scale of self-perceived health. The subscale consists of a single-item rating of health and four additional items reflecting perceived current health, resistance to illness and health outlook. Individual item responses range from 1-5. To score, select items (1, 3, and 5) are recoded so that higher scores indicate better health. The 5 items are then summed and transformed to a 0-100 scale with higher scores reflecting better health.
Change in physical health as assessed by the Pain Intensity scale | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  This consists of one item assessing pain intensity/severity rated on a 11-point scale ranging from 0 (no pain) to 10 (pain so severe you couldn't stand it), higher score indicting worse pain
Change in physical health as assessed by the Interference scale | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  This is a 1 item questionnaire that is scored on a linear scale from 0 (no interference)-10 (extreme interference), higher score indicting worse outcome
Change in physical health as assessed by the SCI Secondary Conditions Scale (SCI-SCS) | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  This is a 16 item questionnaire and each item scores range from 0 (not experienced or insignificant problem) to 3 (significant or chronic problem). Items are summed with a potential score range of 0-48 with higher scores reflecting more severe secondary health conditions.
Change in psychological health and wellbeing as assessed by the Patient Health Questionaire-8 (PHQ-8) | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  This is an 8 item questionnaire and each is scored from 0(not at all) to 3(nearly every day), for a maximum score of 24 higher score indicating worse outcome
Change in psychological health and wellbeing as assessed by the Generalized Anxiety Disorder (GAD-2) scale | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  This is a 2 item questionnaire and each is scored from 0(not at all) to 3(nearly every day), for a maximum score of 6 higher score indicating worse outcome
Change in psychological health and wellbeing as assessed by the 4-itemPerceived Stress Scale (PSS) | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  This is a 4 item questionnaire and questions 1 and 4 are scored from 0(never) to 4(very often) , and questions 2 and 3 are scored from 0(very often) to 4 (never) for a maximum score of 16 higher score indicating worse outcome
Change in psychological health and wellbeing as assessed by the SCI-Qol Positive Affect and Well-being Scale | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  This is a 10 item questionnaire, and each is scored from from 1 (never) to 5 (always). Items are summed to create a raw score. Raw scores are then converted to an IRT-based T-score using provided look-up tables. T-scores range from 26.7 to 68.6 with higher scores representing more positive affect and well-being.
Change in psychological health and wellbeing as assessed by the Diener Satisfaction with Life Scale (SWLS) | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  This is a 4 item questionnaire and each is scored on a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). Scores are summed resulting in a scale score ranging from 4 to 28 with higher scores representing greater life satisfaction.
Change in social health as assessed by the UCLA Loneliness scale | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  This is a 3 item questionnaire and each is scored from 1(hardly ever) to 3(often) for a maximum score of 9 higher score indicating worse outcome
Change in social health as assessed by the Spinal Cord Injury - Quality of Life Scale (SCI-QOL) Satisfaction with Participation Scale | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  This is a 10 item questionnaire and each is scored from 1(not at all) to 5(very much ) with the scale direction depending on whether the item is positively or negatively worded. Item scores are summed to create a raw score which is then converted to an IRT-based T-score using look-up tables. T-scores range from 28.3 to 60.5 with higher scores representing more satisfaction with social roles and activities.

SECONDARY OUTCOMES:
Change in self efficacy as assessed by the Generalized Self-Efficacy Scale (GSES) | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  This is a 10 item questionnaire and each is scored from 1(not at all true) to 4(exactly true), for a maximum score of 40 , higher number indicating better outcome
Change in self efficacy as assessed by the University of Washington Self-efficacy Scale(UW-SES) | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  This is a 6 item questionnaire and each is scored from 1(not at all) to 5(completely) for a maximum score of 30, higher score indicating better outcome
Change in health behaviors/behavioral symptoms as assessed by the Health Promoting Lifestyle Profile-II (HPLP-II) | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  This is a 52 item questionnaire and each is scored from 1(never) to 4(routinely).Items are summed and divided by 52, resulting in a scale score reflecting the average score across all items. This score can range from 1-4, with higher scores reflecting more engagement in health promoting behaviors and practices.
Change in health behaviors/behavioral symptoms as assessed by the SCI-specific Health Behavior Questionnaire (HBQ) | Baseline, end of intervention (8 weeks after baseline), follow up (4 months after end of intervention )
  This is a 22 item questionnaire with each health behavior item scored from 0 (never) to 3 (always) for a maximum score of 66, higher score indicating better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Susan Robinson-Whelen, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- TIRR Memorial Hermann Spinal Cord Injury and Disability Research Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No